CLINICAL TRIAL: NCT06201780
Title: Assessment of Serum Levels of Janus Kinase 1 and 2 in Patients With Cholinergic Urticaria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Elsayed Mohamed, Resident-Dermatology department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-23-12-07MS
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Cholinergic Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases group (Active Comparator): group of cases with cholinergic urticaria
  Interventions: Diagnostic Test: serum levels of Janus Kinase 1and 2
- control group (Active Comparator): control group not have cholinergic urticaria
  Interventions: Diagnostic Test: serum levels of Janus Kinase 1and 2

INTERVENTIONS:
Diagnostic Test: serum levels of Janus Kinase 1and 2 — assessment of serum levels of Janus Kinase 1and 2 by ELISA

SUMMARY:
Cholinergic Urticaria (CholU) is as a subtype of CIndU caused by an increase in the core body temperature, such as to activate the sweating reflex. It can occur in response to physical exercise, hot bathing and/or emotional stress. Clinically it appears as pinpointing and highly pruritic wheals with surrounding erythema, CholU can be accompanied by severe symptoms such as angioedema, respiratory symptoms or anaphylaxi CholU is frequently associated with atopic dermatitis (AD) The JAK-STAT is a mast cell (MC) signaling pathway activated downstream of IgE and IL-3 with important roles in MC homeostasis via regulation of proliferation, survival, and release of mediators. JAK-STAT activation is associated with polarization toward Th2, B cell isotype switching to IgE production, and IgE-dependent degranulation and cytokine release .

Because both IL-4 and IL-13 use the IL-4Rα as a receptor component, these cytokines activate any common signaling pathways. Both of these cytokines use Janus kinases (JAKs) to initiate signaling and activate signal transducer and activator of transcription-6 (STAT6), which is a transcription factor required for many of their biologic functions.

The non-receptor protein tyrosine kinases JAK1 and JAK3 associate with the IL-4Rα and γC, respectively. The binding of IL-4 to its receptor induces the transphosphorylation of JAK1 and JAK3, an event that activates these kinases and thereby initiates the early events of signal transduction .

ELIGIBILITY:
Inclusion Criteria:

* The study will include 45 adult patients complaining of CholU as well as 45 healthy controls.

Exclusion Criteria:

* Patients with one or more of the following criteria will be excluded:

  * Pregnancy and lactation.
  * Patients with systemic diseases especially those with autoimmune diseases and infections.
  * Patients with skin diseases.
  * Patients on medications such as: antibiotics, non-steroidal anti-inflammatory drugs, angiotensin-converting enzyme inhibitors, anticonvulsants, penicillin, combined oral contraceptives.
  * Patient refusal

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
serum levels of janus kinase 1 | 1 year
  assessment of serum levels of janus kinase 1

SECONDARY OUTCOMES:
serum levels of janus kinase 2 | 1 year
  assessment of serum levels of janus kinase 2

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Altrichter S, Koch K, Church MK, Maurer M. Atopic predisposition in cholinergic urticaria patients and its implications. J Eur Acad Dermatol Venereol. 2016 Dec;30(12):2060-2065. doi: 10.1111/jdv.13765. Epub 2016 Jun 21. PMID 27324252
- [Background] Altrichter S, Salow J, Ardelean E, Church MK, Werner A, Maurer M. Development of a standardized pulse-controlled ergometry test for diagnosing and investigating cholinergic urticaria. J Dermatol Sci. 2014 Aug;75(2):88-93. doi: 10.1016/j.jdermsci.2014.04.007. Epub 2014 May 1. PMID 24837213
- [Background] Burchett JR, Dailey JM, Kee SA, Pryor DT, Kotha A, Kankaria RA, Straus DB, Ryan JJ. Targeting Mast Cells in Allergic Disease: Current Therapies and Drug Repurposing. Cells. 2022 Sep 27;11(19):3031. doi: 10.3390/cells11193031. PMID 36230993
- [Background] Fricke J, Avila G, Keller T, Weller K, Lau S, Maurer M, Zuberbier T, Keil T. Prevalence of chronic urticaria in children and adults across the globe: Systematic review with meta-analysis. Allergy. 2020 Feb;75(2):423-432. doi: 10.1111/all.14037. Epub 2019 Oct 11. PMID 31494963